CLINICAL TRIAL: NCT03102567
Title: Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Effect of Aging of Multiple Oral Doses of GLPG1205 in Healthy Male Subjects
Brief Title: This is a Study to Evaluate the Effect of Aging of Multiple Doses of GLPG1205 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1205-CL-105
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Healthy; Elderly
MeSH Terms: interventions — GLPG1205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GLPG1205 50mg q.d. (Experimental): oral hard gelatin capsules with 50 mg GLPG1205 for q.d. administration - compared to placebo
  Interventions: Drug: GLPG1205 50mg q.d.
- placebo (Placebo Comparator): oral hard gelatin capsules containing placebo for q.d. administration
  Interventions: Drug: Placebo oral capsule
- GLPG1205 250 mg loading and 50mg q.d. maintenance (Experimental): open label - oral hard gelatin capsules with 50 mg GLPG1205 for one time 250 mg loading dose and subsequent 50mg q.d. administration
  Interventions: Drug: GLPG1205 250 loading dose and 50mg q.d. maintenance dose

INTERVENTIONS:
Drug: GLPG1205 50mg q.d. — oral gelatin capsule containing 50mg GLPG1205 for q.d. administration - compared to placebo
  Arms: GLPG1205 50mg q.d.
Drug: Placebo oral capsule — oral gelatin capsule containing placebo to match study arm 1 - q.d. administration
  Arms: placebo
Drug: GLPG1205 250 loading dose and 50mg q.d. maintenance dose — Open label - oral gelatin capsule containing 50mg GLPG1205 for one time 250mg loading dose and subsequent q.d. administration
  Arms: GLPG1205 250 mg loading and 50mg q.d. maintenance

SUMMARY:
This study is a Phase I, single-center, randomized, double-blind, placebo-controlled study to evaluate the effect of aging on safety, tolerability and PK of multiple oral doses of GLPG1205 in healthy male subjects.

The study will comprise of 2 parts, a first part to investigate the effect of aging and a second part to investigate the effect of a loading dose.

DETAILED DESCRIPTION:
In Part 1, a total of 24 healthy male subjects matched for weight will be divided into 3 age groups:

* Cohort A: 8 subjects aged 65 to 74 years, inclusive
* Cohort B: 8 subjects aged ≥ 75 years (1:1 weight matched with subjects of Cohort A [±5 kg])
* Cohort C: 8 subjects aged between 18-50 years, inclusive (1:1 weight matched with subjects of Cohort A [±5 kg])

Each cohort will be randomized 3:1 to active (6 subjects) and placebo (2 subjects) treatment respectively. Weight matched subjects in Cohorts B and C will be assigned to active treatment and placebo accordingly. Cohorts A and C will be dosed with 50 mg q.d. GLPG1205 for 14 days.

In the open-label Part 2, an additional cohort of 8 subjects aged 65-74 years (Cohort D) will be included to characterize the PK profile after a loading dose followed by multiple doses of GLPG1205 q.d. for 13 days. A 250 mg loading dose will be administered on Day 1 followed by 50 mg q.d. from Day 2 to Day 14.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged over 18 years
2. Able and willing to sign the ICF.
3. Able and willing to comply with the requirements of the study.
4. Body Mass Index (BMI) between 18 and 30 kg/m² inclusive.
5. Weight between 60 and 90 kg, inclusive (Cohort A only).
6. Considered by the Investigator to be in good health.
7. Discontinuation of all medications with the exception of occasional paracetamol
8. Have a creatinine clearance (estimated by Cockroft-Gault equation) > 80 mL/min for subjects aged up to 50 years in cohort C and > 60 mL/min for subjects of 65 years and over in cohorts A, B and D.
9. A non-smoker and not using any nicotine-containing products .
10. Negative tests for drug screen, alcohol screen, and cotinine screen.
11. Male subjects and their female partners of child-bearing potential must agree to use a highly effective method of contraception.

Exclusion Criteria:

1. Known hypersensitivity to GLPG1205 or excipients of the formulation. A history of significant allergic reaction to any drug, such as anaphylaxis requiring hospitalization.
2. Positive serology for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
3. Clinically significant illness in the 12 weeks prior to study screening.
4. Current or sequelae of gastrointestinal, liver or kidney disease or any other condition that might interfere with absorption, distribution, metabolism or excretion of drugs.
5. History of malignancy in the last 5 years.
6. Clinically significant abnormalities on ECG of rhythm or conduction
7. Clinically significant abnormalities detected on physical examination or vital signs.
8. Clinically significant abnormalities detected on laboratory safety testing
9. Significant blood loss, including blood donation of > 450 mL, or receiving a blood transfusion or blood product in the 12 weeks prior to study screening.
10. Active drug or alcohol abuse within 2 years prior to study screening.
11. Consumption of large quantities of caffeinated coffee or tea (> 6 cups/day), or equivalent. The consumption of alcohol, methyl-xanthine-containing beverages or foods (e.g., coffee, tea cocoa, cola and chocolate), quinine (e.g., tonic water), grapefruit or grapefruit juice, Seville oranges and poppy seeds within 48 h of study medication administration until the end of the dosing period.
12. Concurrent or recent participation in an investigational medicinal research study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Difference between the number of healthy male subjects from different age groups and placebo subjects with adverse events | From screening until the final follow up visit (day 35)
  to assess safety and tolerability in the first placebo controlled part of the study
Difference between the number of healthy male subjects from different age groups and placebo subjects with abnormal laboratory evaluations | From screening until the final follow up visit (day 35)
  to assess safety and tolerability in the first placebo controlled part of the study
Difference between the number of healthy male subjects from different age groups and placebo subjects with abnormal vital signs | From screening until the final follow up visit (day 35)
  to assess safety and tolerability in the first placebo controlled part of the study
Difference between the number of healthy male subjects from different age groups and placebo subjects with abnormal ECG | From screening until the final follow up visit (day 35)
  to assess safety and tolerability in the first placebo controlled part of the study
Difference between the number of healthy male subjects from different age groups and placebo subjects with abnormal physical examination | From screening until the final follow up visit (day 35)
  to assess safety and tolerability in the first placebo controlled part of the study
Difference between healthy male subjects of different age groups of Cmax of GLPG1205 | From day 1 pre-dose until the final follow up visit (day 35)
  To assess PK of GLPG1205 in the first part of the study with different age groups
Difference between healthy male subjects of different age groups of tmax of GLPG1205 | From day 1 pre-dose until the final follow up visit (day 35)
  To assess PK of GLPG1205 in the first part of the study with different age groups
Difference between healthy male subjects of different age groups of AUC0-t of GLPG1205 | From day 1 pre-dose until the final follow up visit (day 35)
  To assess PK of GLPG1205 in the first part of the study with different age groups
Difference between healthy male subjects of different age groups of apparent terminal half-life (t1/2) of GLPG1205 | From day 1 pre-dose until the final follow up visit (day 35)
  To assess PK of GLPG1205 in the first part of the study with different age groups
Assessment of Cmax of GLPG1205 in subjects having received a loading dose of 250mg and subsequent 50mg q.d. maintenance dose | From day 1 pre-dose until the final follow up visit (day 35)
  In the open label (part 2) of the study
Assessment of tmax of GLPG1205 in subjects having received a loading dose of 250mg and subsequent 50mg q.d. maintenance dose | From day 1 pre-dose until the final follow up visit (day 35)
  In the open label (part 2) of the study
Assessment of AUC0-t of GLPG1205 in subjects having received a loading dose of 250mg and subsequent 50mg q.d. maintenance dose | From day 1 pre-dose until the final follow up visit (day 35)
  In the open label (part 2) of the study
Assessment of t1/2 of GLPG1205 in subjects having received a loading dose of 250mg and subsequent 50mg q.d. maintenance dose | From day 1 pre-dose until the final follow up visit (day 35)
  In the open label (part 2) of the study

SECONDARY OUTCOMES:
Assessment of creatinine clearance in healthy elderly subjects | From screening until the final follow up visit (day 35)
  To assess renal function in healthy elderly subjects

CONTACTS AND LOCATIONS:
Overall Officials: Helen Timis, MBChB MICR, Study Director — Galapagos NV
Locations (1):
- SGS clinical pharmacology unit, Antwerp, Belgium